CLINICAL TRIAL: NCT07374744
Title: The Effect Of An Interactive Video-Based Self-Management Education On Glycemic Control, Self-Management and Empowerment İn Individuals With Type 2 Diabetes: A Parallel-Group, Single-Blind, Randomized Controlled Trial
Brief Title: Effect of Interactive Video-Based Self-Management Education in Adults With Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, Associate professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AİBÜ-SBF-IOB-2026
Record Dates: First submitted 2026-01-09; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Outpatient
Keywords: type 2 diabetes mellitus; self management; video recording; education; nursing; empowerment; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Empowerment

STUDY DESIGN:
Intervention Model Description: This study is designed as a parallel-group, single-blind, randomized controlled interventional trial. Eligible adults with type 2 diabetes will be randomly assigned in a 1:1 ratio to either the intervention or control group. Block randomization with a fixed block size of six will be used to ensure balanced group allocation throughout the study period. The randomization sequence will be generated using a computer-based random number system by an independent individual who is not involved in participant recruitment, intervention delivery, or outcome assessment.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study uses a single-blind design. Due to the nature of the intervention, the researcher delivering the intervention cannot be blinded. However, participants will not be informed whether they are assigned to the intervention or control group during data collection. To ensure blinding during data analysis, all study data will be coded using non-identifiable group labels (e.g., Group A/B or Group 1/2). The coded dataset will be provided to an independent statistician, who will be blinded to group allocation during statistical analysis and reporting. This approach is intended to minimize bias and ensure objectivity in outcome evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Nursing Care (Active Comparator)
  Interventions: Behavioral: Standard Nursing Care
- Interactive video training (Experimental)
  Interventions: Behavioral: Interactive video training; Behavioral: Standard Nursing Care

INTERVENTIONS:
Behavioral: Interactive video training — The intervention is designed to promote active learning through decision-making, question-answer interactions, and scenario-based navigation within the video content. The education program is based on the AADE7 Self-Care Behaviors framework and covers healthy coping, healthy eating, physical activity, medication use, monitoring, risk reduction, and problem-solving. Videos are structured around real-life scenarios, performed by an actor portraying a patient, and each video lasts approximately 5-10 minutes. Participants will access the web-based videos via their personal smartphones and will be given one month to complete all content, with unlimited viewing allowed. Engagement will be monitored weekly, and reminders will be provided if no viewing occurs for one week. Interactive elements include embedded questions, feedback videos, and informational prompts. Participant satisfaction will be assessed at the 3-month follow-up.
  Other Names: Interactive video education
  Arms: Interactive video training
Behavioral: Standard Nursing Care — Standard nursing care is routinely provided at the outpatient clinic by a diabetes nurse educator in accordance with established institutional clinical protocols and educational practices. This care consists of face-to-face verbal education delivered during routine follow-up visits. Educational content generally includes core components of diabetes management, such as treatment approaches, self-monitoring of blood glucose, nutrition planning, physical activity recommendations, prevention of acute complications-particularly hypoglycemia-and daily self-care practices. Follow-up visits typically involve reviewing blood glucose records, assessing clinical status, and reinforcing self-management behaviors based on individual needs.

SUMMARY:
This study aims to evaluate the effectiveness of an interactive video-based self-management education program for adults with type 2 diabetes. The education program is designed to support individuals in managing their daily diabetes care and improving their blood glucose control. Participants in this study will be adults diagnosed with type 2 diabetes who are receiving outpatient care. Eligible participants will be randomly assigned to either an intervention group or a control group. Participants in the intervention group will receive an interactive video-based education program developed according to the AADE7 Self-Care Behaviors framework. The videos are based on real-life scenarios and encourage active participation and decision-making. Participants in the control group will receive standard diabetes care. The study will assess changes in blood glucose control, diabetes self-management behaviors, and empowerment levels over the study period. Data will be collected using clinical measurements and questionnaires. Participation in this study is voluntary. The results of this study may contribute to improving diabetes education practices and supporting patient-centered care in clinical settings.

DETAILED DESCRIPTION:
This doctoral thesis study is designed as a parallel-group, single-blind, randomized controlled interventional trial aimed at evaluating the effects of an interactive video-based self-management education program on glycemic control, self-management behaviors, and empowerment in individuals with type 2 diabetes. To ensure methodological transparency and adherence to established scientific reporting standards, the detailed study protocol is planned to be published as a separate scientific article.

Eligible adults with type 2 diabetes will be randomly assigned in a 1:1 ratio to either the intervention or control group. Block randomization with a fixed block size of six will be used to maintain balanced group allocation throughout the study period. The randomization sequence will be generated using a computer-based random number system by an independent individual who is not involved in participant recruitment, intervention delivery, or outcome assessment.

Prior to the main trial, a pilot study will be conducted to assess the acceptability and usability of the developed interactive video-based education program. Findings from the pilot study will be used solely to refine the intervention content and research procedures and will not be included in the sample or final analyses of the main trial. The results of the pilot study are also planned to be reported in a separate scientific publication.

Participants assigned to the intervention group will receive an interactive video-based diabetes self-management education program developed in accordance with the American Association of Diabetes Educators' AADE7 Self-Care Behaviors framework. The educational content will be structured around scenario-based representations of self-care behaviors that individuals with diabetes are expected to perform in their daily lives. The scenarios will be enacted by an individual assuming the role of a patient and will realistically reflect situations commonly encountered in everyday life. Each educational video will have an approximate duration of 5-10 minutes.

The video-based intervention will address the following AADE7 domains: Healthy Coping, Healthy Eating, Being Active, Taking Medication, Monitoring, Reducing Risk, and Problem Solving. Content validity will be established through expert review, with the scenarios evaluated by 10 experts experienced in nursing and internal medicine. Revisions will be made based on expert feedback, and the appropriateness of the educational materials will be assessed using the Davis technique. The finalized scenarios will subsequently be produced as educational videos.

The videos will be converted into an interactive format by incorporating elements such as question-and-answer segments, fill-in-the-blank activities, pop-up informational screens, and highlighted content areas. When participants provide incorrect responses to interactive questions, an explanatory video segment presenting the correct answer will be displayed, with the aim of supporting active learning and enhancing knowledge retention.

Participants in the control group will continue to receive standard routine care. Baseline assessments will be conducted prior to group allocation, and outcome measures will be evaluated at baseline and follow-up to assess changes in glycemic control, diabetes self-management, empowerment, and quality of life. In addition, participants' satisfaction with the educational materials will be assessed at the 3-month follow-up using the Satisfaction Evaluation Form.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years (Mumcu & İnkaya, 2022).
* Able to read, write, understand, and speak Turkish.
* Diagnosed with type 2 diabetes for at least one year (Onyia et al., 2023; Shahshahani et al., 2023).
* Receiving oral antidiabetic agents and/or insulin therapy (Mikhael et al., 2019).
* Having an HbA1c level >7% in at least one measurement within the last 3 months (Hu et al., 2023; Lee et al., 2020; Asmat et al., 2023; TEMD, 2024).
* Volunteering to participate in the study.
* Owning a personal device (e.g., smartphone) capable of playing interactive videos.
* Having the ability to use a smartphone capable of playing interactive videos, which will be assessed by observing the participant using an interactive video -not related to the study intervention.
* Owning a smartphone with an active internet data plan.
* Being able to attend scheduled follow-up visits at the frequency required for study measurements.
* Having a body mass index (BMI) ≥18.5 kg/m² (Lee et al., 2022).
* Not following a vegan or vegetarian diet (Dening et al., 2023).
* Having hemoglobin levels within normal ranges (women: 12-16 g/dL; men: 14-18 g/dL) (Billett, 1990).

Exclusion Criteria:

* Having previously received video-based diabetes education.
* Currently using or having previously used a video-based tool or program supporting type 2 diabetes management.
* Having severe visual, auditory, cognitive impairments, or physical disabilities that may interfere with participation.
* Being hospitalized as an inpatient during the intervention period.
* Being pregnant, planning pregnancy within the next 6 months, or becoming pregnant during the study.
* Breastfeeding during the study period (due to potential dietary restrictions).
* Using any weight-loss medication or supportive pharmacological agent.
* Having a diagnosis of sickle cell anemia or being diagnosed during the study period (TEMD, 2024, p.18; Eyth et al., 2025).
* Receiving hemodialysis, having experienced recent bleeding or blood transfusion, or receiving erythropoietin therapy (TEMD, 2024, p.18; Eyth et al., 2025).
* Having a diagnosed psychiatric disorder (e.g., major depressive disorder, bipolar disorder, schizophrenia).
* Participating in another diabetes-related intervention or program during the study period.
* Using an insulin pump (Lee et al., 2022).
* Managing diabetes with nutrition therapy alone without pharmacological treatment.
* Following a diet prescribed and supervised by a dietitian due to another medical condition or surgical procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The Comprehensive Diabetes Self-Management Scale (CDSMS) | Baseline (prior to intervention) and at 3-month follow-up
  CDSMS is a patient-centered instrument developed to assess self-management behaviors in individuals with diabetes. The scale evaluates key domains of diabetes self-care, including healthy eating, physical activity, medication adherence, blood glucose monitoring, problem-solving, risk reduction, and healthy coping with stress.The CDSMS consists of 14 items (26 questions) with scores ranging from 0 to 4.The total score reflects overall diabetes self-management ability. The scale has demonstrated acceptable internal consistency (Cronbach's alpha=.70-.73) and has been validated for use in the Turkish population. Higher CDSMS scores are associated with better glycemic control, as indicated by HbA1c levels. In the ROC analysis, HbA1c ≤6.50 indicated good glycemic control and >6.50 poor control. Scores below 21 were associated with poor glycemic control. The total CDSMS score is the sum of the seven domain scores and ranges from 0 to 28, with higher scores indicating better self-management.
Hba1c | Baseline (prior to intervention) and at 3-month follow-up
  HbA1c will be used to assess glycemic control. Predefined HbA1c thresholds will be applied for descriptive and interpretive purposes, with lower values indicating better glycemic control and higher values indicating poorer control.
Diabetes Empowerment Scale (DES) | Baseline (prior to intervention) and at 3-month follow-up
  The Diabetes Empowerment Scale (DES) is a validated and reliable self-report scale developed to assess the levels of psychosocial empowerment and self-efficacy in individuals with diabetes regarding diabetes management. The scale consists of three sub-dimensions: management of psychosocial aspects of diabetes, level of dissatisfaction and readiness for change, and setting and achieving diabetes goals. Items are scored from 1 to 5, and sub-dimension and total scores are calculated by averaging the relevant items. Each sub-dimension and total score ranges from 1 to 5. Lower scores indicate lower levels of psychosocial competence and empowerment related to diabetes, while higher scores indicate higher levels of empowerment.
Estimated average glucose (ADAG) | Baseline (prior to intervention) and at 3-month follow-up
  Glycemic control will be evaluated using estimated average glucose (ADAG), which represents mean blood glucose over the previous 2-3 months and is calculated from HbA1c using the formula:
  ADAG (mg/dL) = (28.7 × HbA1c) - 46.7.
Fasting plasma glucose (FPG) | Baseline (prior to intervention) and at 3-month follow-up
  Fasting plasma glucose (FPG) will be used to assess glycemic control and is defined as the plasma glucose concentration measured after at least 8 hours of overnight fasting.

SECONDARY OUTCOMES:
SF-12 Health Survey (Secondary Outcome) | Baseline (prior to intervention) and at 3-month follow-up
  The SF-12 Health Survey is a validated generic instrument developed to assess health-related quality of life over the previous four weeks, independent of age or disease group. The questionnaire consists of 12 items covering eight health domains and generates two summary scores: the Physical Component Summary (PCS-12) and the Mental Component Summary (MCS-12). PCS-12 reflects general health, physical functioning, physical role, and bodily pain, while MCS-12 represents social functioning, emotional role, mental health, and vitality. Scores range from 0 to 100, with higher scores indicating better health-related quality of life. The Turkish version of the SF-12 has demonstrated acceptable reliability for both physical and mental component scores. A high score on the scale indicates that the individual is in good health.

OTHER OUTCOMES:
Other outcomes- Blood pressure | Baseline (prior to intervention) and at 3-month follow-up
  Blood pressure will be measured in mmHg after a period of rest to assess cardiovascular risk as part of diabetes management.
Other outcomes- Body weight | Baseline (prior to intervention) and at 3-month follow-up
  Body weight will be measured in kilograms using a calibrated scale to evaluate changes in overall body mass related to diabetes management.
Other outcomes- Waist circumference | Baseline (prior to intervention) and at 3-month follow-up
  Waist circumference will be measured in centimeters at the midpoint between the lowest rib and the iliac crest to assess central adiposity associated with metabolic risk in diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided